CLINICAL TRIAL: NCT01255488
Title: Family Nurse Practitioner Perception of Journal Abstract Usefulness in Clinical Decision-making: a Randomized Controlled Trial
Brief Title: Research Abstract Usefulness in Clinical Decision-making
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Ronald W. Gimbel, PhD, Uniformed Services University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R02930-S2
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-11

CONDITIONS: Clinical Decision-making
Keywords: Search engine; Clinical decision-making; Research abstracts; Full-text manuscripts; Family Nurse Practitioners

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- EBN-Search (without full-text manuscripts) (Experimental): In the intervention arm research subjects will be provided access to EBN-Search (a fictitious search engine) with nine abstracts relating to the clinical case but no full-text manuscripts.
  Interventions: Behavioral: Access to EBN-Search (without full-text manuscripts)
- EBN-Search (with full text manuscripts) (Active Comparator): Research subjects will be exposed to 9 abstracts and corresponding full-text manuscripts related to the simulated clinical encounter.
  Interventions: Behavioral: Access to EBN-Search (without full-text manuscripts)

INTERVENTIONS:
Behavioral: Access to EBN-Search (without full-text manuscripts) — Family nurse practitioner access to EBN-Search without availability of full-text manuscripts.
  Other Names: Research abstracts; Full-text manuscripts

SUMMARY:
To better understand the extent to which family nurse practitioners (FNPs) might use research abstracts in shaping their clinical decision-making under simulated conditions. A secondary point is to examine if and how FNPs might use full-text manuscripts (associated with the abstracts) if made available to them.

DETAILED DESCRIPTION:
The study will recruit the approximate 25 - 1st year and 25 - 2nd year family nurse practitioner students of the Graduate School of Nursing. After being presented an overview of the study and informed consent document, those electing to participate will draw a sealed envelope indicating whether they are assigned to group A (intervention group) or group B (control group). The participant will proceed to the associated room, be provided a brief clinical case (appropriate to their training), an iPad device with pre-loaded EBN-Search engine, and a questionnaire. The EBN-Search engine for the intervention group will include 9 research abstracts associated to the case. The EBN-Search for the control group will include both the research abstracts and full-text versions of the manuscripts. The participants will be provided 20 minutes to complete the questionnaire using the information available to them. The questionnaire will require the participant to indicate treatment plan, respond to questions regarding the usefulness of research abstracts, questions regarding the usefulness of full-text (control group only) and recommendations on improving EBN-Search.

ELIGIBILITY:
Inclusion Criteria:

* Matriculated family nurse practitioner graduate students of USUHS 2010/2011 academic year

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-03 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Measure of perception of abstract usefulness in clinical decision-making | Immediate post-experiment
  At conclusion of the simulated exercise subjects will complete a data collection instrument indicating their perception of abstract usefulness in their clinical decision-making.

SECONDARY OUTCOMES:
Use of full-text manuscripts when available in simulated clinical encounter | During experiment
  For those subjects with ready access to full-text manuscripts (n=25) during the simulated clinical encounter, we will measure how often they are accessed by the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W. Gimbel, PhD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Uniformed Services University, Bethesda, Maryland, United States